CLINICAL TRIAL: NCT00623987
Title: Absence of Residual Vein Thrombosis After an Episode of Unprovoked Deep Vein Thrombosis: Short-Term Anticoagulation is Safe.
Brief Title: Absence of Residual Vein Thrombosis Permits to Withdrawn Oral Anticoagulants
Acronym: Exten-DACUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico (Other)
Responsible Party: Sergio Siragusa, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0036/99
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Deep Vein Thrombosis
Keywords: Residual vein thrombosis; Optimal duration; Oral anticoagulants
MeSH Terms: conditions — Venous Thrombosis | interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): warfarin treatment
  Interventions: Drug: warfarin accordingly INR value
- B (No Intervention): withholding warfarin therapy

INTERVENTIONS:
Drug: warfarin accordingly INR value — warfarin accordingly to INR value between 2.0-3.0
  Other Names: warfarin
  Arms: A

SUMMARY:
Background. The optimal duration of oral anticoagulant treatment in patients with idiopathic Deep Vein Thrombosis (DVT)of the lower limbs is still uncertain. Residual Vein Thrombosis (RVT) has been found able to establish the patient' risk for recurrent thrombotic events. In the present study we conducted a RVT-based therapeutic strategy, withholding OAT after 3 months in patients without RVT while continuing anticoagulants for at least additional 9 months in those in whom RVT persists.

Methods Patients with a first episode of symptomatic unprovoked proximal Vein Thrombosis (VT) were given Oral Anticoagulant Treatment (OAT) for 3 months. Residual Vein Thrombosis (RVT), ultrasonographically-detected, will be then assessed. Patients without RVT did not continue OAT (Group B), whereas those with RVT will continue OAT for at least additional 9 months. Patients were followed-up prospectively focusing on the study outcomes: occurrence of recurrent venous thromboembolism and major bleeding over a period of at least 12 months after OAT discontinuation.

DETAILED DESCRIPTION:
INTRODUCTION Long-term anticoagulant treatment with adjusted doses of vitamin K antagonists is highly effective in preventing recurrent events after a first episode of unprovoked Venous ThromboEmbolism (VTE), even if the optimal duration of this therapy is still uncertain. Since the risk of recurrency is greatest in the first year after the initial thrombotic episode and gradually diminishes thereafter, the benefit of an extended course of anticoagulant treatment may be offset over time by the persisting risk of clinically important bleeding.

A potential clinically relevant approach for establishing the optimal duration of Oral AntCoagulant Therapy (OAT) is that of predicting the individual risk for thrombotic recurrency after the index Deep Vein Thrombosis (DVT). Although the current scheme for establishing the duration of OAT is based on the nature of index DVT (idiopathic or provoked), some new data starting to select other parameters to optimize this decision. Recently, the use of D-dimer has been proven to be effective for selecting OAC duration; however, this investigation evaluated only patients with idiopathic DVT and, moreover, the use of D-dimer can not be easily handle by most of Institutions.

In earlier prospective studies conducted in patients with symptomatic DVT, the presence of a residual thrombus was associated with an increased risk of thrombotic recurrencies either in idiopathic or provoked venous thrombosis. Interestingly, recurrent events occurred not only in the previously affected veins but also in other sites, thus suggesting that Residual Vein Thrombosis (RVT) may express a pro-thrombotic status. Based on these findings, the detection of RVT may be, therefore, of help in establishing the duration of anticoagulation. Recently, we have conducted a randomized, prospective, follow-up study in patients with a first episode of symptomatic DVT treated with OAT for 3 months in whom OAT duration was based upon RVT findings. In patients without RVT, the risk of recurrent DVT was low even if the treatment was stopped after only 3 months.

To further confirm our preliminary data and to enforce the safety of withholding OAT after 3 months in patients without RVT, we conducted a prospective study in patients with idiopathic DVT of the lower limbs.

METHODS Study patients. Patients with a first episode of documented unprovoked and provoked proximal DVT will be eligible for the study if they had completed at least three months of OAT (target INR 2.5, range 2.0-3.0). Unprovoked DVTs are defined as thrombotic episodes occurred in apparently healthy individuals. Patients with active cancer, limited life expectancy, antiphospholipid antibody syndrome, or an other known thrombophilic status (such as antithrombin deficiency), serious liver disease, those who lived too far from the center will be excluded from the study. The study has been approved by the institutional review boards of all participating centers. All enrolled patients will provide written informed consent.

Study Design. This is a multicenter prospective study in patients with a first episode of symptomatic proximal DVT detected by Compression UltraSonography (C-US) and receiving OAT [warfarin (Coumadin, Bristol Myers Squibb) for 3 months. At this time, subjects who agreed to participate have a physical examination to assess baseline clinical conditions and to exclude contraindications. C-US of the proximal deep vein system in both legs will be performed, measuring the diameters of any detectable thrombus in the Common Femoral Vein (CFV) and Popliteal Veins (PV). Images will be obtained in transverse section only. Lumen compressibility will be then evaluated on CFV and PV by gentle pressure of the probe, as previously described. Briefly, the major and the minor diameters of the vein segment are measured and recorded before and after compression. C-US findings are scored as "absence of RVT" when residual thrombus occupied, at maximum compressibility, less than 40% of the vein area. Patients without RVT will not continue anticoagulation (Group B), whereas those with RVT will continue OAT (INR 2.0-3.0) for at least additional 9 months.

Study outcomes and Follow-up. From the assignment visit, patients will be followed up for at least one year after OAT discontinuation; during the follow-up period, patients will be contacted by the clinical centers every 3 months. C-US will be performed only when recurrent symptomatic DVT is suspected. The study outcome is the composite of confirmed recurrent venous thromboembolism (including DVT and/or fatal or non-fatal pulmonary embolism) and major bleeding events from the index DVT to the last day of follow-up. In cases of suspected DVT recurrence the results of ultrasonography will be compared with the previous examination. A diagnosis of recurrent venous thrombosis is made if a previously fully compressible segment (contralateral or ipsilateral) became incompressible. In absence of a previous normal C-US, DVT recurrence is diagnosed if a previously non-occlusive thrombus shifted to occlusive thrombus, provided the vein area before compression had increased > 4 mm); in undetermined cases, contrast venography was performed. In patients with suspected pulmonary embolism, diagnosis of recurrence is based on objective algorithms using clinical probability, ventilation-perfusion lung scanning/helical computed tomography, compression ultrasonography and/or D-dimer if indicated. The diagnosis of clinically relevant haemorrhage will be made in case of decrease of haemoglobin levels > 2.0 gr/dl, retroperitoneal, intracranial or life-threatening. Patients has been instructed to contact the clinical center immediately if symptoms developed suggestive of venous thromboembolism or bleeding. All suspected outcome events and all deaths will be evaluated by a central adjudication committee whose members were unaware of the name of the subject, the enrolling center, the C-US findings and the assigned group.

Statistical analysis. Baseline differences between groups will be assessed by the chi-square test (Yates' correction) for categorical variables and t-test or Mann-Withney U test for continuous variables, as appropriate. Data will be analyzed on intention-to-treat basis. Kaplan-Meier survival curves are plotted to estimate the cumulative incidence of symptomatic recurrent venous thromboembolism and major bleeding. Patients who during the study will develop clinical conditions interfering with the study outcomes (such as ischemic heart disease, cancer, stroke, superficial vein thrombosis, etc) and left the assigned group will be regularly followed-up and included in analysis. Hazard ratios and their 95 percent confidence intervals will be calculated using the Cox's proportional hazards model. The data will be analyzed using the Prism statistical software package (Version 3.0, GraphPad Software Incorporated, San Diego, CA) and the SPSS statistical package (Version 14.0, SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* First episode of unprovoked proximal DVT of the lower limbs and treated for 3 month with oral anticoagulants

Exclusion Criteria:

* Active cancer,
* Limited life expectancy,
* Antiphospholipid antibody syndrome, or an other known thrombophilic status (such as antithrombin deficiency),
* Serious liver disease,
* Pregnancy
* Conditions requiring anticoagulation (atrial fibrillation, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 1999-06; Primary Completion 2006-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Recurrent Venous Thromboembolism | for the entire study

SECONDARY OUTCOMES:
major and minor haemorrhage, death | for the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Siragusa, MD, Study Chair — University Hospital of Palermo
Locations (1):
- Sergio Siragusa, Palermo, Italy

REFERENCES:
- [Derived] Siragusa S, Malato A, Saccullo G, Iorio A, Di Ianni M, Caracciolo C, Coco LL, Raso S, Santoro M, Guarneri FP, Tuttolomondo A, Pinto A, Pepe I, Casuccio A, Abbadessa V, Licata G, Battista Rini G, Mariani G, Di Fede G. Residual vein thrombosis for assessing duration of anticoagulation after unprovoked deep vein thrombosis of the lower limbs: the extended DACUS study. Am J Hematol. 2011 Nov;86(11):914-7. doi: 10.1002/ajh.22156. Epub 2011 Sep 22. PMID 21953853